CLINICAL TRIAL: NCT04554420
Title: Promoting Youth Mental Health in Inequitable Contexts: Applying Participatory Action Research
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Given recruitment challenges for youth focus groups, we are currently finalizing the creation of the intervention based on the focus groups. We plan to submit for new grant funding to implement a different intervention at a future date.
Sponsor: Charles Drew University of Medicine and Science (Other)
Collaborators: Los Angeles County Department of Public Health (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: U54MD007598 (NIH)
Record Dates: First submitted 2020-09-02; First posted 2020-09-18 (Actual); Last update posted 2024-04-02 (Actual); Status verified 2023-11

CONDITIONS: Youth Participatory Action Research; Youth Mental Health; Health Equity

STUDY DESIGN:
Intervention Model Description: Participants (youth) will receive intervention (mental health curriculum) and a pre-intervention and post-intervention survey will be used to evaluate the intervention. Additionally, a set of focus groups will be conducted post-intervention to assess the feasibility, implementation process, and youth responsiveness. No control condition will be used for this pilot intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Youth Participatory Action Research-Mental Health Curriculum (Experimental): Youth will be engaged with youth participatory approaches in learning about the intersection of mental health and systemic/community level issues.
  Interventions: Behavioral: Youth Participatory Action Research-Mental Health Curriculum

INTERVENTIONS:
Behavioral: Youth Participatory Action Research-Mental Health Curriculum — The mental health curriculum will focus on enhancing the knowledge, critical consciousness (i.e., exploration of systemic/racial problems), research self-efficacy, and other skills of youth to integrate their lived experiences and identity to learning about the intersection of system and community level issues in mental health. Activities will center on participatory action approaches to engaging youth in culturally/community responsive ways.

SUMMARY:
The current study addresses the gap in equity in mental health education for adolescents of color in South Los Angeles. Particularly, the focus is on developing, testing and evaluating the feasibility and youth responsiveness of a curriculum reflecting the main principles/concepts of the framework of "Youth Participatory Action Research" and general mental health outcomes for adolescents living in a context of poverty and significant inequities.

DETAILED DESCRIPTION:
In order to effectively prevent mental distress and promote well-being for youth of color in urban contexts with significant health inequities and mental health stigma, more innovative and participatory models are critical. Youth participatory action research (YPAR), is a framework outlining engagement of youth with researchers more equitably as co-constructors of knowledge and promoting positive development of core competencies in youth to foster their growth as change agents. YPAR is especially valuable for youth of color, to build competencies (e.g., critical consciousness, research and advocacy skills) critical for tackling health inequities and systems change. The proposed study will be conducted in partnership with the Community Healing and Trauma Prevention Center (CHTPC), a community grass roots organization of the Los Angeles County Department of Public Health, charged with designing educational and creative spaces for prevention and healing of trauma in the community, with youth positive development as one of its key priorities. Guided by YPAR, this mixed-method, pre-post evaluation study will develop a YPAR-Mental Health (MH) curriculum and evaluate its feasibility, youth responsiveness, and association with positive youth developmental outcomes related to YPAR and mental health with youth of color (ages 14-17) from high schools in South Los Angeles (SPA-6). The study will comprise two phases: Phase 1 - Development and Refinement of YPAR-MH Curriculum, and Phase 2 - Pilot Testing, Implementation and Evaluation of YPAR-MH Curriculum. During phase 1, a team of the PI, CDU graduate students, King/Drew Magnet High School students, and CHTPC staff will develop the curriculum. Input for refinement of the curriculum will be offered by a team of youth experts, including: a) community youth advocates, b) clinical psychologist with youth mental health expertise, and c) community psychologist with YPAR expertise. A set of four focus groups will be conducted with youth (4-6 youth per focus group, 14-17 years of age) to further improve the curriculum to assure "youth responsiveness".

During phase 2, a total of 20 youth will participate in the pilot testing of the YPAR-MH curriculum. After further refining the curriculum given lessons learned from the pilot testing, a total of 50 youth will participate in the finalized curriculum implementation. A pre-post curriculum survey will be conducted for all youth. Additionally, a set of four focus groups with youth participating in the finalized curriculum will be conducted to evaluate their qualitative experiences, satisfaction with curriculum, and learning of curriculum material. There are two specific aims, objectives and hypotheses which will be tested:

Specific Aim 1: To develop and refine a YPAR-MH curriculum, guided by youth community, research, and clinical experts. Four focus groups will be conducted with a maximum total of 24 youth to assess the youth responsiveness of the curriculum. A qualitative thematic analysis of the focus group data will be conducted and the findings will be used to further refine the curriculum.

Specific Aim 2: To finalize and evaluate the curriculum with a pre-post survey and focus groups.

Objective 1: Conduct pilot testing of curriculum with 20 youth to further improve and finalize curriculum.

Objective 2: Implement the finalized curriculum with 50 youth and examine the change in youth outcomes pre to post curriculum based on evaluation survey and four focus groups.

Hypothesis 2a: Youth will experience a significant positive improvement from pre to post curriculum for YPAR related outcomes: critical consciousness, research self-efficacy, and ethnic/racial identity.

Hypothesis 2b: Youth will experience a modest positive improvement from pre to post curriculum for mental health related outcomes: anxiety and depression, stress, and resilience.

ELIGIBILITY:
Inclusion Criteria:

* High school age youth, 14-17 years old
* Youth living in South Los Angeles

Exclusion Criteria:

* Not meeting the age range of 14-17 years old
* Youth not living in South Los Angeles

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2024-02 (Estimated); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Critical Consciousness Scale - Assessing change from pre-intervention to immediately post-intervention | Measure will be implemented pre-intervention and immediately post-intervention
  Measure assesses capacity to critically analyze socio-political conditions, endorsement of social equity, and action to change perceived inequities; Subscale/Sample Item/Number of Items: a) Critical reflection perceived inequality: "Poor children have fewer chances to get a good high school education" (n=8), b) Critical reflection egalitarianism: "Group equality should be our ideal" (n=5), c) Critical action socio-political participation: "Participate in a discussion about a social or political issue (n=9); 6 point Likert- type (Strongly disagree to Strongly agree)
Research Self-Efficacy - Assessing change from pre-intervention to immediately post-intervention | Measure will be implemented pre-intervention and immediately post-intervention
  Measure assesses perceived self-efficacy to conduct and analyze research; Sample item/Number of items: "I believe I can master research related knowledge" (n=4); 5 point Likert-type (Strongly disagree to Strongly Agree)
Multigroup Ethnic Identity Measure - Assessing change from pre-intervention to immediately post-intervention | Measure will be implemented pre-intervention and immediately post-intervention
  Measure assesses multiple dimensions of ethnic/racial identity, including the following; Subscale/Sample items/Number of items: a) Ethnic behaviors: "I participate in cultural practices of my own group" (n=4), b) Affirmation and belonging: "I have a lot of pride in my ethnic group" (n=6), c) Ethnic identity achievement: "In order to learn more about my group, I have often talked to other people about my group" (n=4); 4 point Likert-type (Strongly disagree to Strongly agree)
Revised Child Anxiety and Depression Scale-Short Version - Assessing change from pre-intervention to immediately post-intervention | Measure will be implemented pre-intervention and immediately post-intervention
  Measure assesses anxiety and depression in the general population/non-clinical of youth; Subscale/Sample items/Number of items: a) Anxiety: "Worries about things" (n=15), b) Depression: "Feels worthless" (n=10); 4 Likert-type (Never to Always)
Adolescent Distress-Eustress Scale - Assessing change from pre-intervention to immediately post-intervention | Measure will be implemented pre-intervention and immediately post-intervention
  Measure assesses distress (negative stress) and eustress (positive stress) in adolescents; Subscale/Sample items/Number of items: a) Distress: "I felt overwhelmed" (n=5), b) Eustress: "I felt motivated" (n=5); 5 point Likert-type (Not like me to Very much like me)
Child and Youth Resilience Measure-28 - Assessing change from pre-intervention to immediately post-intervention | Measure will be implemented pre-intervention and immediately post-intervention
  Measure assesses resilience in youth; Subscale/Sample items/Number of items: a) Individual: "I cooperate with people around me" (n=11), b) Caregiving: "My caregivers watch me closely" (n=7), c) Contextual: "I am treated fairly in my community" (n=10); 5 point Likert-type (Does not describe me at all to Describes me a lot)

CONTACTS AND LOCATIONS:
Overall Officials: Noe R Chavez, PhD, Principal Investigator — Charles Drew University of Medicine and Science

IPD SHARING:
Plan to Share IPD: No